CLINICAL TRIAL: NCT03833674
Title: Acute Intermittent Hypoxia and Respiratory Strength Training to Improve Breathing Function After Spinal Cord Injury
Brief Title: FLO2 for Recovery After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802672; W81XWH-18-1-0718 (Other Grant/Funding Number: US Deptartment of Defense)
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: acute intermittent hypoxia (AIH); spinal neuroplasticity; motor function; respiratory strength training; respiration; breathing; plasticity
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: Participants will complete a battery of clinical assessments and 4 randomly ordered intervention and testing blocks. Blocks 1, 2 and 3 include a 5 day intervention (e.g., dAIH and/or respiratory training) or sham protocol, followed by a 3-week washout period, with follow up measurements at 1 day, 3 days and 1 week post-intervention. The final block includes a 5-day protocol followed by 1-day, 3-day and 1-week post-tests.
Masking Description: Participants and the clinical evaluator will be informed of possible interventions but will be blinded to the gas mixture (hypoxic vs normoxic air) used during each AIH intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with incomplete SCI (Experimental): Adults with chronic, incomplete SCI who have >20% impairment in respiratory function, who will complete a battery of clinical assessments and 4 randomly ordered intervention and testing blocks (Daily AIH Block, Sham dAIH Block, Respiratory Strength Training Block and AIH + Strength Training Block).
  Interventions: Other: Daily AIH Block; Other: Sham dAIH Block; Other: Respiratory Strength Training Block; Other: AIH + Strength Training Block

INTERVENTIONS:
Other: Daily AIH Block — Daily sessions of AIH (dAIH) with use of short episodes of low oxygen (9% O2)
  Other Names: dAIH Block
Other: Sham dAIH Block — Daily sessions of sham dAIH which includes breathing room air (21% O2)
Other: Respiratory Strength Training Block — Respiratory strength training using a hand-held device that resists inspiration or expiration.
Other: AIH + Strength Training Block — AIH followed by respiratory strength training.

SUMMARY:
Acute intermittent hypoxia (AIH) involves short (~1-2min) bouts of breathing low oxygen air to stimulate spinal neuroplasticity. Studies in rodents and humans indicate that AIH improves motor function after spinal cord injury (SCI). This study will use a double blind, cross-over design to test if the combination of AIH and respiratory strength training improves breathing function more than either approach alone in adults with chronic SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) disrupts neural pathways to respiratory motor neurons, causing muscle paralysis and decreased breathing capacity. Since respiratory impairment is the major cause of illness and death with SCI, it is critical to devise new strategies to restore breathing function.

Repetitive exposure to brief episodes of low oxygen (acute intermittent hypoxia or AIH) has demonstrated to increase respiratory function in humans with chronic SCI. Additionally pre-clinical studies demonstrate that AIH-induced functional benefits are enhanced by combining AIH with task-specific training. The investigator's central hypothesis is that combined daily AIH (dAIH) and respiratory strength training will elicit greater and more sustained gains in respiratory function than either treatment alone in people with chronic SCI.

This study is a double-blind, randomized, cross-over design where participants will complete 4 random-ordered blocks, consisting of a 5-day intervention followed by a 3-week washout period, during which 1-day, 3-day, and 1-week post-tests will be conducted. Participants will include 53 adults with chronic, incomplete SCI with >20% respiratory impairment based on maximal inspiratory or expiratory pressure generation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic incomplete SCI for ≥ 1 year at or below C-1 to T-12
* Incomplete SCI based on residual sensory and motor function below the level of the injury or injury classification of B, C, D at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI

-OR-

Chronic complete SCI for ≥ 1 year at or below C-4 to T-12

* Complete SCI based on the absence of residual sensory or motor function below the level of injury or injury classification of A at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI.
* Medically stable with clearance from physician
* SCI due to non-progressive etiology
* >20% impairment in maximal inspiratory or expiratory pressure generation, relative to established normative values.

Exclusion Criteria:

* Current diagnosis of an additional neurologic condition such as multiple sclerosis, Parkinson's disease, stroke, or brain injury
* Presence of unstable or uncontrolled medical conditions such as cardiovascular disease, myocardial infarction, <1 year lung disease, infections, hypertension, heterotopic ossification.
* Severe neuropathic pain
* Known pregnancy
* Severe recurrent autonomic dysreflexia
* History of seizure disorder < 1 year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in maximal inspiratory pressure | Baseline, Day 1, Day 6, Day 8, Day 15
  Maximal inspiratory pressure is a non-invasive measure of the maximal force achieved when breathing in against an occluded airway.
Change in maximal expiratory pressure | Baseline, Day 1, Day 6, Day 8, Day 15
  Maximal expiratory pressure is a non-invasive measure of the maximal force generated when breathing out against an occluded airway.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, PT, PhD, Principal Investigator — University of Florida; Gordon Mitchell, PhD, Principal Investigator — University of Florida
Locations (1):
- Brooks Rehabilitation Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welch JF, Vose AK, Cavka K, Brunetti G, DeMark LA, Snyder H, Wauneka CN, Tonuzi G, Nair J, Mitchell GS, Fox EJ. Cardiorespiratory Responses to Acute Intermittent Hypoxia in Humans With Chronic Spinal Cord Injury. J Neurotrauma. 2024 Sep;41(17-18):2114-2124. doi: 10.1089/neu.2023.0353. Epub 2024 Apr 18. PMID 38468543